CLINICAL TRIAL: NCT05502796
Title: Natural History and Pathogenesis of Alopecia in Children and Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000827; 000827-AR
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Hair Loss
Keywords: Skin Conditions; Autoimmune Disease; Natural History
MeSH Terms: conditions — Alopecia; Skin Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Male and female ages 2-45 years old

SUMMARY:
Background:

Alopecia is the loss of hair or lack of hair growth. It is often related to an immune disorder that disrupts the growth of hair. Hair loss can affect a person s physical and mental health. The causes of alopecia are not well understood. This natural history study will examine causes of alopecia so better treatments can be developed.

Objective:

To learn why some people have alopecia. This study will look at factors related to genes, the immune system, and the bacteria, viruses, and fungi that live on the skin.

Eligibility:

People aged 2 years and older with immune-mediated alopecia that affects 50% of their scalp hair.

Design:

Participants will have at least 1 visit to the clinic. Some will have follow-up visits once a year for up to 5 years. Each visit will last 2 to 4 hours.

Participants will have a physical exam. They will have blood drawn from a vein. They will answer questions about the medications they take, their allergies, and their family history. Photographs of their skin and scalp will be taken. Soft cotton swabs will be rubbed on their skin to pick up organisms that live there.

Two pieces of skin from the scalp will be cut away. The pieces will be no more than a quarter of an inch in size. The area will first be numbed with an injectable anesthetic. The wound will be closed with stitches or gel foam. The biopsy is optional in children younger than 12.

Participants will take a questionnaire about how hair loss affects their quality of life.

DETAILED DESCRIPTION:
Study Description:

This is a study to detail the characteristics (genetic, immunologic, biological and demographic) of individuals who present in childhood and adulthood with alopecia and how alopecia impacts skin and systemic symptoms.

Objectives:

Primary objective: Comprehensively evaluate patients with immune mediated alopecia from clinical, microbiome, immunologic and genetic standpoint to understand the factors that contribute to clinical phenotypes.

Secondary objective: To follow patients with immune-mediated alopecia to see how disease impacts local skin microbiome, immune system changes and autoimmune and other comorbidities.

Tertiary objectives: To develop prognostic biomarkers that help predict the risk of severity and progression in patients with alopecia.

Endpoints:

1. Record demographics including age, sex, age of onset, severity of disease based on clinical examination, concomitant autoimmune disease, personal history of other medical disease including anxiety and depression, family history of autoimmune and medical disease
2. Whole genome sequencing to identify variations in the protein-coding region of any gene that may be disease causing
3. Assess peripheral blood and local scalp skin to assess immunogenicity of disease by using leukocyte subset analysis using flow cytometry, markers of disease using cytokine signaling assays, and single cell RNA sequencing
4. Define skin microbiome using sequencing at baseline and with time.
5. Identify potential biomarkers of disease progression or severity that may impact therapeutic choices

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with study procedures including skin biopsy of the scalp (except in those under the age of 12 years) and availability for the duration of the study
2. Willing to avoid using antibacterial cleansers for 1 week prior to sampling
3. Male or female, aged 2 years and older
4. Clinical Diagnosis of immune- mediated alopecia
5. Ability of subject or Parent/legal guardian to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Non-immune mediated alopecia including androgenetic alopecia, radiation induced alopecia, trauma induced alopecia, chemotherapy induced alopecia
2. Concomitant medical, surgical, or other conditions for which adequate facilities or funds are not available to support their care at the NIH.
3. Any other co-existing condition/circumstances that would make a subject unsuitable to participate in the study, as deemed by the investigators.
4. Pregnant women

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who present in childhood and adulthood with alopecia.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Describe the natural history of alopecia based on demographics, whole exome sequencing, and microbiome and immunologic signals | 5 years

SECONDARY OUTCOMES:
Explore immune system, microbiome signals during flares and quiescence as well as during therapy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi H Kong, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000827-AR.html